CLINICAL TRIAL: NCT02947880
Title: Evaluation of the Efficiency of Treatment by BUMETANIDE on Autistic Children With a Known Ethiology : Multicenter and Double Blind-study With Randomized Parallel Group, Against Placebo.
Brief Title: Evaluation of the Efficiency of Treatment by BUMETANIDE on Autistic Children With a Known Ethiology
Acronym: BUMAUTEP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the recently feasibility study shows that the number of patients is insufficient in the centers
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: I14039
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2017-08

CONDITIONS: Autistic Disorder
Keywords: autism, Bumetanide
MeSH Terms: conditions — Autistic Disorder | interventions — Bumetanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bumetanide group (Experimental): During 3 months in the double blind, the patient will receive the experimental treatment. For the patient of 25kg and more the bumetanide is used at the posology of 1mg in the morning and 1mg in the evening, for patient under 25kg the posology is 0.5mg in the morning and 0.5mg in the evening.
  After the 3 months in the double blind trial (bumetanide versus placebo), all the patient will receive (in the open phase of the trial) the bumetanide during 3 months with the posology fitting with their weights.
  Interventions: Drug: Bumetanide
- Placebo group (Placebo Comparator): During 3 months in the double blind, the patient will receive the placebo. For the patient of 25kg and more the bumetanide is used at the posology of 1mg in the morning and 1mg in the evening, for patient under 25kg the posology is 0.5mg in the morning and 0.5mg in the evening.
  After the 3 months in the double blind trial (bumetanide versus placebo), all the patient will receive (in the open phase of the trial) the bumetanide during 3 months with the posology fitting with their weights.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bumetanide — For the patient of 25kg and more the bumetanide is used at the posology of 1mg in the morning and 1mg in the evening, for patient under 25kg the posology is 0.5mg in the morning and 0.5mg in the evening.
  Arms: Bumetanide group
Drug: Placebo — For the patient of 25kg and more the placebo is used at the posology of 1mg in the morning and 1mg in the evening, for patient under 25kg the posology is 0.5mg in the morning and 0.5mg in the evening.
  Arms: Placebo group

SUMMARY:
During a previous therapeutic trial, investigators showed that the bumetanide improved significantly autism. This trial showed that a therapeutic response was obtained in 75% of cases.

These first results were reinforced by a study led with adult patients for whom the eye tracking measurements as well as the functional MRI showed a diminution of the response time and a modification (amplification) of the cerebral response during an emotions recognition test.

Finally, investigators confirmed the physiological mechanism behind the action of the bumetanide in a study in two mouse models of autism.

ELIGIBILITY:
Inclusion Criteria:

* Children and teenager from age 5 to age 17, with a diagnosis of typical autism or Asperger syndrome according to the criteria of diagnosis of the WHO's classification (CIM-10),
* With a known etiology,
* Patients for whom the CARS results are strictly Superior or equal to 30,
* Of whom the parents have given their free, informed and written consent,
* Affiliated or beneficiary of the French social security.

Exclusion Criteria:

* Patients under treatment by inlet diuretic either at the time of the study or before,
* Patients with electrolytic disorders,
* Patients with a known hypersensitivity to sulfa drugs,
* Patients with a hepatic or renal failure,
* Patients with an epilepsy not controlled by a treatment (comitial crisis in the past 6 month at the time the trial starts despite a treatment),
* Patients under treatment by psychotropic exception made of the melatonin,
* Allergy to the bumetanide or one of its excipients,
* Patient under a treatment by lithium, diphemanil, erythromycin IV, halofantrine, pentamidine, sultopride, vincamine, aminoglycoside,
* Pregnant and lactating women.

Secondary exclusion criteria:

* QT prolongation noticed on the ECG at Day0,
* Anomaly on the biological check up (Day 0) made before including the patient that would contraindicated the prescription of bumetanide,
* Patients for whom the CARS results are strictly inferior to 30.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change (evolution) between day 0 and day 99 of the result of the scale CARS (Childhood Autism Rating Scale). | Day 0 and Day 99

SECONDARY OUTCOMES:
CARS (Childhood Autism Rating Scale) between D0 and D99 and between D99 and D190 which will be describe by etiology | Day 0, Day 99 and Day 190